CLINICAL TRIAL: NCT02499172
Title: Follow-up of Pregnant Women After a Mass Vaccination of Oral Cholera Vaccine
Brief Title: Follow-up of Pregnant Women After a Mass Vaccination of Oral Cholera Vaccine (ShancholTM) in Nsanje Malawi
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial reason
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Ministry of Health, Malawi (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00006369
Record Dates: First submitted 2015-07-07; First posted 2015-07-16 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Miscarriage; Stillbirth; Cholera
Keywords: Adverse pregnancy outcome
MeSH Terms: conditions — Abortion, Spontaneous; Stillbirth; Cholera | interventions — shanchol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Cohort 1: Women who were pregnant and received at least one dose of ShancholTM during the mass OCV vaccination campaign.
  Interventions: Biological: Shanchol
- Cohort 2 (No Intervention): Cohort 2: Women who received at least one dose and who became pregnant after the mass vaccination campaign; hence their fetuses were not exposed to the vaccine.
- Cohort 3 (No Intervention): Cohort 3: Women who were pregnant in Chikwawa District at the time of the vaccination campaign in Nsanje District, but who did not receive the vaccine during the campaign.
- Cohort 4 (No Intervention): Cohort 4: Women who become pregnant in Chikwawa District after the vaccination campaign in Nsanje District, and who did not receive the vaccine during the campaign.

INTERVENTIONS:
Biological: Shanchol
  Arms: Cohort 1

SUMMARY:
This study, to be carried out immediately following an emergency, reactive cholera vaccination campaign in Nsanje District, Malawi, will be a cohort study to estimate the safety of killed oral cholera vaccine (OCV), in pregnant women as measured by ShancholTM, on pregnancy outcomes and birth defects. While limited evidence which suggests that the vaccine is safe in pregnant women, this setting will allow investigators to answer this question in a community where more than 100,000 people will receive vaccine with no restrictions on pregnancy status. In past cholera vaccine campaigns including clinical trials, pregnant women were excluded due to lack of safety data. However, in this campaign, the decision by the Ministry of Health is that the benefits of offering vaccine to all individuals regardless of pregnancy status far outweigh any theoretical risk. Here the investigators specifically propose to:

Specific Objective 1: To conduct surveillance of pregnant women to detect adverse pregnancy outcomes within communities in Nsanje District, Malawi that received oral cholera vaccine in a reactive vaccination campaign that started on 30 March 2015. Through household surveying and enrollment of pregnant women with monthly follow-up visits, the investigators will determine the cumulative incidence of adverse pregnancy outcomes among vaccinated and unvaccinated women in Nsanje and Chikwawa Districts, Malawi.

Specific Objective 2: To compare the cumulative incidence of pregnancy loss (miscarriage and stillbirth) of women who received oral cholera vaccine while they were pregnant to women who were vaccinated and became pregnant after the end of the final round of vaccination in Nsanje and Chikwawa Districts, Malawi.

Specific Objective 3: To compare the incidence of newborn malformations in a cohort of infants that had fetal exposure to oral cholera vaccine compared to those without such exposure in Nsanje and Chikwawa Districts, Malawi.

DETAILED DESCRIPTION:
Although there are good reasons for women of reproductive age to participate in interventions that prevent cholera, cholera vaccination programs and studies have generally excluded pregnant women since there is little specific information on the safety of the vaccine during pregnancy. However, there are several biological reasons why inactivated OCVs are unlikely to have a harmful effect on fetal development. First, the bacteria in the vaccine are killed and do not replicate. Second, the vaccine antigens act locally on the gastrointestinal mucosa, are not absorbed, and do not enter the maternal or fetal circulation. Finally, the vaccines do not trigger systemic reactions (e.g., fever) associated with miscarriage in early pregnancy.According to the latest WHO position paper in relation to OCV, vaccination in countries where cholera is endemic may include groups that are particularly vulnerable to the severe forms of cholera, and for whom the vaccines are not contraindicated, such as pregnant women and HIV-infected individuals.

While the World Health Organization (WHO) recommends vaccination for pregnant women, the package inserts for Dukoral® and ShancholTM are more cautious and suggests that the vaccines are not recommended for use in pregnant women. Even so, the ShancholTM package insert states that, "Administration of ShancholTM to pregnant women may be considered after careful evaluation of the benefits and risks in case of a medical emergency or an epidemic". In the most recent results published in 2012, pregnant women inadvertently vaccinated with Dukoral® during the mass vaccination campaign in Zanzibar in 2009 did not experience any harmful effects. On the other hand, there is no information on the safety of ShancholTM vaccine in pregnant women. New evidence is needed to inform decisions on the true safety of this vaccine in pregnancy. If it is safe, this vaccine will be a valuable tool in reducing the burden of cholera in a population that disproportionately suffers from this disease.

On January 13, 2015, the President of the Republic of Malawi declared a state of disaster following the persistent rains that resulted in floods affecting 15 of the 28 districts in the country. The first confirmed case of cholera was reported in Malawi on February 11, 2015. As of 4 March 2015, Malawi had registered 72 cases with 2 deaths. To stop the outbreak of cholera, a cholera vaccination campaign program was carried out between 30 March 2015 and May 3 2015 targeting the camps and the nearby communities in Nsanje District. This campaign provided two doses of vaccine to all age eligible people irrespective of pregnancy status. This study is designed to do a follow-up of only the pregnant women aiming at the following objectives:

Specific Objective: To conduct surveillance of pregnant women to detect adverse pregnancy outcomes within communities in Nsanje District, Malawi that received oral cholera vaccine in a reactive vaccination campaign that started on 30 March 2015. Through household surveying and enrollment of pregnant women with monthly follow-up visits, the investigators will determine the cumulative incidence of adverse pregnancy outcomes among vaccinated and unvaccinated women in Nsanje and Chikwawa Districts, Malawi.

ELIGIBILITY:
Inclusion criteria:

* Women aged 15-49 years old at time of consent (all cohorts)
* Urine sample provided if pregnancy test required (Not required if experienced delivery outcome between March 30 and enrollment date, OR visibly pregnant AND has due date indicated in Health Passport) (all cohorts)
* Received at least one dose of OCV in 2015 (must be verified with OCV Vaccination Card) (Cohorts 1 & 2)
* Estimated last menstruation at least 3 weeks before the first dose of OCV received (Nsanje) or before March 30, 2015 (Chikwawa) (Cohorts 1 & 3)
* Estimated last menstruation at least 2 weeks after the final dose of OCV received (Nsanje) or after the last day of OCV Round 2 (Chikwawa) (Cohorts 2 & 4)
* Residing in Nsanje or Chikwawa Districts since the first day of the vaccination campaign (30 March 2015) (Cohorts 2 & 3)
* Provides informed consent (with additional consent by the parent or legal guardian for unmarried <18 years old) (All Cohorts)

Exclusion criteria:

* Received at least one dose of OCV in 2015 (Cohorts 3 & 4)
* An otherwise eligible pregnant women who is unable to be contacted after the second attempt within 48 hours after the first attempt to enroll (All cohorts)

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2758 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10-30 (Actual); Study Completion 2016-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Ali M, Nelson A, Luquero FJ, Azman AS, Debes AK, M'bang'ombe MM, Seyama L, Kachale E, Zuze K, Malichi D, Zulu F, Msyamboza KP, Kabuluzi S, Sack DA. Safety of a killed oral cholera vaccine (Shanchol) in pregnant women in Malawi: an observational cohort study. Lancet Infect Dis. 2017 May;17(5):538-544. doi: 10.1016/S1473-3099(16)30523-0. Epub 2017 Feb 2. PMID 28161570

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Cohort 1: Women who were pregnant and received at least one dose of ShancholTM during the mass OCV vaccination campaign.
  Shanchol: Oral cholera vaccine
- Cohort 3: Cohort 3: Women who were pregnant in Chikwawa District at the time of the vaccination campaign in Nsanje District, but who did not receive the vaccine during the campaign.
  Non-intervention: Non recipients of the vaccine
- Cohort 2: Cohort 2: Women who were not pregnant and received at least one dose of ShancholTM during the mass OCV vaccination campaign.
  Shanchol: Oral cholera vaccine
- Cohort 4: Cohort 4: Women who were not pregnant and not received any dose of ShancholTM during the mass OCV vaccination campaign.
  Shanchol: Oral cholera vaccine
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 3 | Cohort 2 | Cohort 4
Started | 900 | 899 | 523 | 436
Completed | 835 | 835 | 0 | 0
Not Completed | 65 | 64 | 523 | 436
Not completed — Financial reason | 0 | 0 | 523 | 436
Not completed — Lost to Follow-up | 65 | 64 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 2: Cohort 2: Women who were not pregnant in at the time of the vaccination campaign in Nsanje District, but who did not receive the vaccine during the campaign.
- Cohort 4: Cohort 4: Women from Chikwawa who were not pregnant in at the time of the vaccination campaign in Nsanje District, but who did not receive the vaccine during the campaign.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 3 | Cohort 2 | Cohort 4 | Total
Number analyzed (Participants) | 835 | 835 | 523 | 436 | 2629
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.93 (6.51) | 25.75 (6.81) | 24.24 (6.51) | 25.32 (6.61) | 25.84 (6.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 835 | 835 | 523 | 436 | 2629
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Malawi | 835 | 835 | 523 | 436 | 1670

OUTCOME MEASURES:

1. Primary Outcome: Adverse Pregnancy Outcome
Description: The primary analysis will compare adverse pregnancy outcome (miscarriage and stillbirth) in Cohorts 1 and 3.
Time Frame: Upto 42 weeks from the date of last menstrual period
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Cohort 2: Women who were not pregnant at the time of the vaccination campaign in Nsanje District, but who received receive the vaccine during the campaign.
- Cohort 4: Cohort 4: Women who were not pregnant in Chikwawa District at the time of the vaccination campaign in Nsanje District, but who did not receive the vaccine during the campaign.
Arm/Group | Cohort 1 | Cohort 3 | Cohort 2 | Cohort 4
Number analyzed (Participants) | 835 | 835 | 523 | 436
Participants | 46 | 36 | 19 | 18

ADVERSE EVENTS:
Groups:
- Cohort 2: Cohort 2: Women who were not pregnant at the time of the vaccination campaign in Nsanje District, but who did receive the vaccine during the campaign.
- Cohort 4: Cohort 4: Women who were not pregnant at the time of the vaccination campaign in Nsanje District, but who did not receive the vaccine during the campaign.
Arm/Group | Cohort 1 | Cohort 3 | Cohort 2 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 1/835 | 1/835 | 0/523 | 0/436
Serious Adverse Events (participants affected / at risk) | 0/835 | 0/835 | 0/523 | 0/436
Other Adverse Events (participants affected / at risk) | 0/835 | 0/835 | 0/523 | 0/436

LIMITATIONS AND CAVEATS:
All the participants could not be followed up due to financial reason

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No